CLINICAL TRIAL: NCT00006005
Title: Phase II Study of Thalidomide (NSC #66847) in Patients With Sarcomas of Gynecologic Origin
Brief Title: Thalidomide in Treating Patients With Gynecologic Sarcomas
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: New York University Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000068013; NYGOG-99-001; NCI-314; NYOG-0102-073
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2004-08

CONDITIONS: Endometrial Cancer; Sarcoma
Keywords: stage I uterine sarcoma; stage II uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; recurrent uterine sarcoma; uterine carcinosarcoma; uterine leiomyosarcoma; endometrial stromal sarcoma
MeSH Terms: conditions — Endometrial Neoplasms; Sarcoma; Sarcoma, Endometrial Stromal | interventions — Thalidomide

INTERVENTIONS:
Drug: thalidomide

SUMMARY:
RATIONALE: Thalidomide may stop the growth of gynecologic sarcomas by stopping blood flow to the tumor.

PURPOSE: Phase II trial to study the effectiveness of thalidomide in treating patients who have recurrent or persistent gynecologic sarcomas.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the impact on survival and the antitumor effects of thalidomide in patients with sarcomas or carcinosarcoma (mixed mesodermal tumors) of gynecologic origin.
* Determine the safety and side effect profiles of the target dose of this treatment regimen in this patient population.
* Determine the antiangiogenic and immunologic effects of this treatment regimen in these patients.

OUTLINE: Patients receive oral thalidomide daily. Treatment continues in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed sarcoma or carcinosarcoma (mixed mesodermal tumors) of gynecologic origin not amenable to resection or radiotherapy
* Measurable disease

  * Lesions accurately measured in at least 1 dimension of at least 20 mm in longest diameter with conventional techniques or at least 10 mm with helical CT scan
  * Histologically or cytologically confirmed neoplastic nature if solitary lesion
  * No nonmeasurable disease, defined as:

    * Bone lesions
    * Leptomeningeal disease
    * Ascites
    * Pleural/pericardial effusion
    * Inflammatory breast disease
    * Lymphangitis cutis/pulmonis
    * Unconfirmed abdominal masses not followed by imaging techniques
    * Cystic lesions
* Documented recurrence or persistence following appropriate surgery, radiotherapy, and/or chemotherapy
* Postmenopausal or status post hysterectomy

PATIENT CHARACTERISTICS:

Age:

* Not specified

Performance status:

* ECOG 0-1

Life expectancy:

* Not specified

Hematopoietic:

* Granulocyte count at least 1,000/mm^3
* Platelet count at least 50,000/mm^3

Hepatic:

* Bilirubin normal
* Transaminases less than 2.5 times upper limit of normal

Renal:

* Creatinine less than 1.5 mg/dL

Other:

* No grade 2 or greater peripheral neuropathy
* No medical or social factors that would preclude study, including inability to take oral medication
* No other serious illness requiring immediate therapy
* Not pregnant

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 4 weeks since prior chemotherapy (6 weeks since mitomycin or nitrosoureas)

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics

Other:

* At least 30 days since any prior noncytotoxic experimental antiemetic or antifungal investigational drug

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-09; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Wadler, MD, Study Chair — Weill Medical College of Cornell University
Locations (10):
- United States (10):
  - Cancer Center of Albany Medical Center, Albany, New York
  - North Shore University Hospital, Manhasset, New York
  - St. Vincent's Comprehensive Cancer Center, New York, New York
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - St. Luke's-Roosevelt Hospital Center - Roosevelt Division, New York, New York
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Albert Einstein Clinical Cancer Center, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - University of Wisconsin Comprehensive Cancer Center, Madison, Wisconsin